CLINICAL TRIAL: NCT04727905
Title: Sports Science Institute
Brief Title: The Effect of Supplementing Different Solutions on Firefighters' Simulated Fire Rescue Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, LinYuChih, Principal Investigator, National Taiwan Sport University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB-20-051-A2
Record Dates: First submitted 2021-01-14; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Injury of Multiple Muscles and Tendons at Lower Leg Level
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- energy drink (Experimental): Intake after exercise
  Interventions: Dietary Supplement: energy drink
- Seasoned water (Placebo Comparator): Intake after exercise
  Interventions: Dietary Supplement: energy drink

INTERVENTIONS:
Dietary Supplement: energy drink — The explosive force and muscle endurance of the lower limbs were tested first, and then the special training intervention for fire rescue was performed. Solution supplementation was carried out. The experiment group was divided into the control group and only drank 1 liter of pure water, and the sports drink group supplemented with commercially available sports drinks (using commercially available treasures). Mineral water powder configuration), mint-flavored sports drink group supplemented with mint-flavored commercially available sports drinks (using commercially available treasure mineral water powder configuration plus edible flavor 0.01% menthol)

SUMMARY:
One of the three major tasks of firefighters is disaster rescue, and fire rescue accounts for the majority. They must wear personal protective equipment (PPE) at the fire site during execution. This set of equipment plus other equipment required for rescue will always It weighs up to 40 kg, and the rescue environment is extremely hot and the rescue mission must be carried out in a short time. Under this extremely high pressure, firefighters must have speed, agility, strength and endurance that are different from ordinary people. However, after performing the above fire rescue tasks, firefighters often lose a lot of water; therefore, the purpose of this study is to explore the impact of water and electrolyte supplementation on physical recovery after firefighters perform fire rescue tasks. A total of 24 field firefighters from the Fire Department were research subjects.

In the past research on firefighters, there was no research on the effect of water and electrolyte supplementation on physical recovery after dehydration after performing fire rescue tasks. Therefore, in this study, the body composition was measured before and after the special training of firefighters simulated fire rescue. , Collect venous blood; Replenish electrolytes in sections after training, and take venous blood, urine and saliva for tests at 15, 30 and 60 minutes to analyze relevant values and perform strength tests to observe firefighters The state of physical recovery.

The experiment was divided into three groups. The control group only drank 1 liter of pure water, the sports drink group was supplemented with commercially available sports drinks, and the mint flavored sports drink group was supplemented with mint flavored commercially available sports drinks. Drink 1 liter of liquid within 60 minutes after training; 8 people in each of the 3 groups are randomly assigned. The results of the experiment were analyzed by analysis of variance (ANOVA), and Tukey-Kramer test was used to detect whether there are differences between different treatments, and P<0.05 represents statistical significance.

ELIGIBILITY:
Inclusion Criteria:

- male firefighters aged between 20 and 50

Exclusion Criteria:

* cardiovascular disease hypertension metabolic syndrome glucose-6-acid dehydrogenase deficiency

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Blood biochemical value | one day
  Creatinine
Blood biochemical value | one day
  blood urea nitrogen
Blood biochemical value | one day
  lactate

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided